CLINICAL TRIAL: NCT05813873
Title: The Use of Incentive Spirometry (Triflow) in Patients With Long Covid
Brief Title: The Use of Incentive Spirometry in Adult Patients Hospitalised in a Rehabilitation Center With Long-covid Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Collaborators: Eden Resort Wellness Rehabilitation Center (Unknown)
Responsible Party: Principal Investigator, Marina Kloni, Marina Eleni Kloni, BSc, MSc, MA, European University Cyprus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Triflow
Record Dates: First submitted 2023-04-12; First posted 2023-04-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-03

CONDITIONS: Long COVID
Keywords: Triflow, Incentive Spirometry, Long-covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triflow (Experimental): Use of Triflow device and exercise regime
  Interventions: Other: Triflow
- Control (Active Comparator): Only exercise regime
  Interventions: Other: Control

INTERVENTIONS:
Other: Triflow — Triflow
  Other Names: Triflow and exercise regime
  Arms: Triflow
Other: Control — Exercise
  Other Names: Exercise regime
  Arms: Control

SUMMARY:
The aim of this clinical trial is to investigate the efficacy of Triflow in the rehabilitation of patients with long covid syndrome hospitalised in a rehabilitation center. Participants will be divided into 2 groups and follow their exercise regime until the day they are discharged from the rehabilitation center. The intervention group will participate in a rehabilitation program which includes upper and lower limbs exercises, cycle ergometer, walking and the use of triflow. The control group will participate in the same program but without the Triflow.

DETAILED DESCRIPTION:
Randomised controlled trial with 2 groups:Triflow and exercises (intervention) and exercises (control)

Exercises:Exercises in the bed, chair and standing with/without weights, walking, cycle ergometer, treadmill.

Triflow: 10 breaths in and 10 breaths out.

Both groups will have 1 physiotherapy session per day for 6 days per week from admission to discharge.

Sample size:The sample size is 70. We took into consideration the efficacy of completing the recruitment of patients in time. There few published studies with the use of Triflow as their primary intervention with smaller sample sizes.

Population: Adults with long covid hospitalised in the rehabilitation center

Statistical Analysis: will be done through IBM SPSS Statistics 20 and the level of statistical significance will be (p < 0.05).

From the literature and international guidelines, physiotherapy should be offered to people hospitalized with long-COVID, without any serious risks and offering significant benefit.

ELIGIBILITY:
Inclusion Criteria:

* Adults who were infected with COVID-19 in the last 6 months and were diagnosed with long-covid syndrome
* Patients must be willing to give written consent for participation in the study
* Negative rapid test for COVID-19

Exclusion Criteria:

* History of diseases that do not allow exercise (e.g. unstable cardiac disease)
* Age < 18 years of age
* Significant cognitive and psychiatric impairments (inability to follow simple commands or give consent)
* Lack of will to do the exercises or refuse to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Barthel Index | on admission day
  Measures performance in activities of daily living (eg.stairs, dressing/undressing, washing,eating). Score from 0 to 100, where 0 indicates total dependence and 100 total independence with activities of daily living.
Barthel Index | on discharge day
  Measures performance in activities of daily living (eg.stairs, dressing/undressing, washing,eating). Score from 0 to 100, where 0 indicates total dependence and 100 total independence with activities of daily living.
Dyspnoea (Medical Research Council Dyspnoea Scale) | on admission day
  Assess dyspnoea via MRC dyspnoea scale. The participants grade their dyspnoea on a scale of 1 to 5. The bigger the number, the worse their dyspnoea is
Dyspnoea (Medical Research Council Dyspnoea Scale) | on discharge day
  Assess dyspnoea via MRC dyspnoea scale. The participants grade their dyspnoea on a scale of 1 to 5. The bigger the number, the worse their dyspnoea is
Peak Flow Meter | on admission day
  Assess the respiratory function via peak flow meter. The participants will take a deep breath and blow the air out into the peak flow meter. The higher the score the better their respiratory function is
Peak Flow Meter | on discharge day
  Assess the respiratory function via peak flow meter. The participants will take a deep breath and blow the air out into the peak flow meter. The higher the score the better their respiratory function is

SECONDARY OUTCOMES:
Number of hospitalisation days | on discharge day
  Number of days participants stay in the rehabilitation center
Muscle strength (Hand Grip) | on admission day
  Assess muscle strength for the upper extremities via hand-held dynamometer
Muscle strength (Hand Grip) | on discharge day
  Assess muscle strength for the upper extremities via hand-held dynamometer
Muscle strength and endurance (30 seconds Sit to stand) | on admission day
  Assess muscle strength for the lower extremities and endurance via 30 seconds sit to stand. The participants will have to stand up from a chair without using their arms as many times as they can in 30 seconds. The more times the better their muscle strength and endurance
Muscle strength and endurance (30 seconds Sit to stand) | on discharge day
  Assess muscle strength for the lower extremities and endurance via 30 seconds sit to stand. The participants will have to stand up from a chair without using their arms as many times as they can in 30 seconds. The more times the better their muscle strength and endurance
Balance (Berg Balance) | on admission day
  Assess via Berg Balance Questionnaire, a total of 14 items that asess balance. from 0 to 56, the higher the score the better balance a person has and has a smaller risk for falls.
Balance (Berg Balance) | on discharge day
  Assess via Berg Balance Questionnaire, a total of 14 items that asess balance. from 0 to 56, the higher the score the better balance a person has and has a smaller risk for falls.
Cardiorespiratory fitness (Six minutes walking test) | on admission day
  Assess the cardiorespiratory fitness via 6 minutes walking test. The participants have to walk for 6 mins independently and the distance they cover is measured. The bigger the distance the better cardiorespiratory fitness.
Cardiorespiratory fitness (Six minutes walking test) | on discharge day
  Assess the cardiorespiratory fitness via 6 minutes walking test. The participants have to walk for 6 mins independently and the distance they cover is measured. The bigger the distance the better cardiorespiratory fitness.
Quality of life (EQ-5D-5L) | on admission day
  Assess via EQ-5D-5L questionnaire, it has 6 components (movement,self-care, everyday activities, pain/discomfort, stress/depression, and a scale from 0 to 100 for participants to score how they perceive their health on the day( 0 indicates worst heath and 100 best health)
Quality of life (EQ-5D-5L) | on discharge day
  Assess via EQ-5D-5L questionnaire, it has 6 components (movement,self-care, everyday activities, pain/discomfort, stress/depression, and a scale from 0 to 100 for participants to score how they perceive their health on the day( 0 indicates worst heath and 100 best health)
Fatigue (Multidimensional fatigue inventory) | on admission day
  Assess the feeling of fatigue via Multidimensional fatigue inventory. it has 20 questions with a scale from 1(yes that is true) to 5 (no that is not true)
Fatigue (Multidimensional fatigue inventory) | on discharge day
  Assess the feeling of fatigue via Multidimensional fatigue inventory. it has 20 questions with a scale from 1(yes that is true) to 5 (no that is not true)
Timed up and Go | on admission day
  Assesses mobility and fall risk. Participants have to walk 3m, the shorter the time the better their mobility
Timed up and Go | on discharge day
  Assesses mobility and fall risk. Participants have to walk 3m, the shorter the time the better their mobility

CONTACTS AND LOCATIONS:
Overall Officials: Marina Kloni, Principal Investigator — European University Cyprus
Locations (1):
- Eden Resort Wellness Rehabilitation Center, Larnaca, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basoglu OK, Atasever A, Bacakoglu F. The efficacy of incentive spirometry in patients with COPD. Respirology. 2005 Jun;10(3):349-53. doi: 10.1111/j.1440-1843.2005.00716.x. PMID 15955148
- [Background] Eltorai AEM, Szabo AL, Antoci V Jr, Ventetuolo CE, Elias JA, Daniels AH, Hess DR. Clinical Effectiveness of Incentive Spirometry for the Prevention of Postoperative Pulmonary Complications. Respir Care. 2018 Mar;63(3):347-352. doi: 10.4187/respcare.05679. Epub 2017 Dec 26. PMID 29279365
- [Background] Imamura M, Mirisola AR, Ribeiro FQ, De Pretto LR, Alfieri FM, Delgado VR, Battistella LR. Rehabilitation of patients after COVID-19 recovery: An experience at the Physical and Rehabilitation Medicine Institute and Lucy Montoro Rehabilitation Institute. Clinics (Sao Paulo). 2021 Jun 14;76:e2804. doi: 10.6061/clinics/2021/e2804. eCollection 2021. PMID 34133481
- [Background] Mohamed AA, Alawna M. Role of increasing the aerobic capacity on improving the function of immune and respiratory systems in patients with coronavirus (COVID-19): A review. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):489-496. doi: 10.1016/j.dsx.2020.04.038. Epub 2020 Apr 28. PMID 32388326
- [Background] Seyller H, Gottlieb M, Colla J. A breath of fresh air: The role of incentive spirometry in the treatment of COVID-19. Am J Emerg Med. 2021 Oct;48:369. doi: 10.1016/j.ajem.2021.01.084. Epub 2021 Feb 1. No abstract available. PMID 33558097
- [Background] Siddiq MAB, Rathore FA, Clegg D, Rasker JJ. Pulmonary Rehabilitation in COVID-19 patients: A scoping review of current practice and its application during the pandemic. Turk J Phys Med Rehabil. 2020 Nov 9;66(4):480-494. doi: 10.5606/tftrd.2020.6889. eCollection 2020 Dec. PMID 33364571
- [Background] Spielmanns M, Pekacka-Egli AM, Schoendorf S, Windisch W, Hermann M. Effects of a Comprehensive Pulmonary Rehabilitation in Severe Post-COVID-19 Patients. Int J Environ Res Public Health. 2021 Mar 7;18(5):2695. doi: 10.3390/ijerph18052695. PMID 33800094
- [Background] Zampogna E, Paneroni M, Belli S, Aliani M, Gandolfo A, Visca D, Bellanti MT, Ambrosino N, Vitacca M. Pulmonary Rehabilitation in Patients Recovering from COVID-19. Respiration. 2021;100(5):416-422. doi: 10.1159/000514387. Epub 2021 Mar 30. PMID 33784696
- [Background] Franklin E, Anjum F. Incentive Spirometer and Inspiratory Muscle Training. 2023 Apr 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK572114/ PMID 34283480
- [Background] Restrepo RD, Wettstein R, Wittnebel L, Tracy M. Incentive spirometry: 2011. Respir Care. 2011 Oct;56(10):1600-4. doi: 10.4187/respcare.01471. PMID 22008401
- [Background] Toor H, Kashyap S, Yau A, Simoni M, Farr S, Savla P, Kounang R, Miulli DE. Efficacy of Incentive Spirometer in Increasing Maximum Inspiratory Volume in an Out-Patient Setting. Cureus. 2021 Oct 4;13(10):e18483. doi: 10.7759/cureus.18483. eCollection 2021 Oct. PMID 34754645